CLINICAL TRIAL: NCT00962884
Title: Assessment of Inspiratory Breathing Devices to Improve Orthostatic Tolerance in Neurogenic Orthostatic Hypotension
Brief Title: Breathing Device for Orthostatic Hypotension (OH)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No volunteers were enrolled, study was closed
Sponsor: Alfredo Gamboa (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Alfredo Gamboa, Research Assistant Professor of Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 090600
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Orthostatic Hypotension
Keywords: Orthostatic hypotension; Breathing; Blood pressure; standing
MeSH Terms: conditions — Hypotension, Orthostatic; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITD breathing device (Experimental): Breathing through the Res-Q-Gard ITD device from Advanced Circulatory Systems Inc.
  Interventions: Device: Inspiratory Threshold Device (Res-Q-Gard ITD)
- Sham Device (Sham Comparator): Breathing device similar to active Res-Q-Gard device but with one-way resistance valve removed.
  Interventions: Device: Sham Inspiratory Threshold Device

INTERVENTIONS:
Device: Inspiratory Threshold Device (Res-Q-Gard ITD) — Patient will breathe through this device attached to a mouthpiece during assessment of orthostatic tolerance.
  Other Names: Res-Q-Gard ITD device 7.0 (Ref:12-0463-000)
  Arms: ITD breathing device
Device: Sham Inspiratory Threshold Device — Breathing through device similar to active device but with the one-way threshold valve removed.
  Other Names: Res-Q-Gard device 7.0 (with active valve removed)
  Arms: Sham Device

SUMMARY:
The investigators will test whether breathing through an inspiratory resistance device will improve the ability to be upright and decrease blood pressure drops on standing in patients with orthostatic hypotension.

DETAILED DESCRIPTION:
Orthostatic hypotension is commonly described, especially in an elderly population. Using data from a national hospital inpatient database, Shibao et al. have reported that the annual hospitalization rate for orthostatic hypotension was 233 per 100000 among patients older than 75 years. Orthostatic hypotension is associated with an increased risk of falls, increased risk of coronary heart disease and mortality.

Orthostatic hypotension is defined as a fall in systolic blood pressure of at least 20 mmHg within 3 minutes upon standing 3. Patients with orthostatic hypotension commonly experience lightheadedness or syncope. In normal individuals, changes in posture do not results in significant changes in blood pressure due to physiological compensation for the gravity-mediated pooling of blood in the lower limbs with upright posture. Unfortunately, in patients with impairments of the autonomic nervous system, one or more of these adaptive mechanisms fail, and an orthostatic fall in blood pressure results.

In this pilot study, we will test the hypothesis that breathing through an inspiratory resistance device will improve orthostatic tolerance and reduce orthostatic hypotension in patients with neurogenic orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with neurogenic orthostatic hypotension by the Vanderbilt Autonomic Dysfunction Center
* Decrease in systolic blood pressure ≥ 20 mmHg with position change from supine to standing (10 minutes)
* Evidence of reproducibility suggestive of non-reversible nervous system origin for the orthostatic hypotension
* Age between 18-80 years
* Male and female subjects are eligible
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for orthostatic hypotension (such as acute dehydration)
* Inability to give, or withdrawal of, informed consent
* Pregnant
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Magnitude of drop in Systolic Blood Pressure during head-up tilt | 1 min

SECONDARY OUTCOMES:
"Standing Time" tolerated with systolic blood pressure above 70 mmHg | 10 min (max)
Symptom rating | 10 min (max)
Hemodynamics (non-invasive) | 10 min

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Convertino VA, Ryan KL, Rickards CA, Cooke WH, Idris AH, Metzger A, Holcomb JB, Adams BD, Lurie KG. Inspiratory resistance maintains arterial pressure during central hypovolemia: implications for treatment of patients with severe hemorrhage. Crit Care Med. 2007 Apr;35(4):1145-52. doi: 10.1097/01.CCM.0000259464.83188.2C. PMID 17334239
- [Background] Convertino VA, Ratliff DA, Crissey J, Doerr DF, Idris AH, Lurie KG. Effects of inspiratory impedance on hemodynamic responses to a squat-stand test in human volunteers: implications for treatment of orthostatic hypotension. Eur J Appl Physiol. 2005 Jul;94(4):392-9. doi: 10.1007/s00421-005-1344-1. Epub 2005 Apr 28. PMID 15864634
- [Background] Shibao C, Grijalva CG, Raj SR, Biaggioni I, Griffin MR. Orthostatic hypotension-related hospitalizations in the United States. Am J Med. 2007 Nov;120(11):975-80. doi: 10.1016/j.amjmed.2007.05.009. PMID 17976425
- See also: Vanderbilt Autonomic Dysfunction Center Website — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction